CLINICAL TRIAL: NCT02411695
Title: A Phase 1, Multicenter, Open-label, Dose-Escalation Trial to Assess the Safety, Tolerability and Pharmacokinetics of Oral Brexpiprazole (OPC- 34712) in Adolescents With Schizophrenia
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral Brexpiprazole (OPC- 34712) in Adolescents With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 331-10-233
Record Dates: First submitted 2014-05-30; First posted 2015-04-08 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
Keywords: Adolescent; Otsuka,; Brexpiprazole
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 0.5 mg, Brexpipraxzole (OPC-34712)
  Interventions: Drug: Brexpiprazole (OPC-34712)
- Cohort 2 (Experimental): 1mg, Brexpipraxzole (OPC-34712)
  Interventions: Drug: Brexpiprazole (OPC-34712)
- Cohort 3 (Experimental): 2mg, Brexpipraxzole (OPC-34712)
  Interventions: Drug: Brexpiprazole (OPC-34712)
- Cohort 4 (Experimental): 3 mg, Brexpipraxzole (OPC-34712)
  Interventions: Drug: Brexpiprazole (OPC-34712)
- Cohort 5 (Experimental): 4mg, Brexpipraxzole (OPC-34712)
  Interventions: Drug: Brexpiprazole (OPC-34712)

INTERVENTIONS:
Drug: Brexpiprazole (OPC-34712) — Subjects who are deemed eligible for the trial will be assigned to a dosing cohort and will enter a Dose Titration Phase during which they will receive a starting dose of brexpiprazole for 2 to 10 days based on their assigned titration schedule. The Dose Titration Phase may be extended up to a maximum of 14 days, based on the observed safety and tolerability profile of the previous cohort's Dose Titration Phase. Following the Dose Titration Phase, subjects will enter the Fixed Dose Phase and will be administered the assigned dose for that cohort for 14 days.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of oral brexpipirazole in adolescent subjects with schizophrenia or Other Related Psychiatric Disorders.

DETAILED DESCRIPTION:
Schizophrenia is a severely delibitating mental illness that affects approximately 1% of the world population. The onset of schizophrenia symptoms typically peaks in late adolescence and early adulthood. In a minority of cases, the initial episode may occur during childhood or early adolescence. Patients who experience this "early-onset schizophrenia" exhibit symptoms that are more severe and follow a more chronic course; adolescents with schizophrenia may never achieve full remission of the initial episode. The prognosis for early-onset schizophrenia tends to be poor, and cognitive impairment is greater compared with individuals whose onset of schizophrenia occurs later in life. Several antipsychotics have been investigated for the treatment of adolescent schizophrenia, however, there is a particular challenge because developing bodies are more sensitive to side effects of antipsychotics, particularly with respect to weight gain. In order to enroll a population that includes the younger ages, adolescents with other related psychiatric disorders are also included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 13 to 17 years of age, inclusive, at the time of informed consent.
* Subjects with a current diagnosis of primary schizophrenia spectrum or bipolar spectrum disorder, as defined by DSM-IV-TR criteria, and confirmed by K-SADS-PL.
* No psychiatric hospitalizations within the past 12 weeks.
* Subjects require treatment with antipsychotic medications.
* Subjects who have received previous outpatient antipsychotic treatment at an adequate dose for an adequate duration (at least 6 weeks) and who showed a previous good response to such antipsychotic treatment (other than clozapine) in the last 12 months.
* Subjects with a body weight at Screening greater than or equal to 30 kg.

Exclusion Criteria:

* Sexually active females of childbearing potential and male subjects who are not practicing two different methods of birth control with their partner (or abstinence) during the trial and for 30 days after the last dose of trial medication
* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving trial drug.
* Subjects who have received continuous medication therapy to treat schizophrenia and schizophrenia spectrum diagnosis for less than six months prior to first dose of study medication AND subjects who have received continuous medication therapy to treat bipolar and bipolar spectrum disorder for less than two months in the past three years; or subjects who require more than one antipsychotic..
* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia spectrum , bipolar spectrum, including any Axis I or Axis II (DSM-IV-TR) disorder.
* Subjects with a clinical presentation and/or history of any neurodevelopmental disorder
* Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days.
* Subjects who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any history of myocardial infarction, congestive heart failure, HIV seropositive status/acquired immunodeficiency syndrome, or chronic hepatitis B or C.
* Subjects with IDDM (ie, any subjects using insulin) are excluded. Subjects with non-IDDM may be eligible for the trial if their condition is stable.
* Subjects with epilepsy or a history of seizures.
* Any major surgery or blood transfusion within 30 days prior to first dose of trial medication.
* Subjects with a positive drug screen for cocaine or other illicit drugs, or alcohol are excluded and may not be retested or re-screened.
* Prohibited concomitant medications used within the exclusionary period prior to Day 1 of the Dose Escalation Phase or anticipated need for such medications during the trial.
* Subjects who participated in a clinical trial and were exposed to IMP within the last 30 days or who participated in more than two interventional clinical trials within the past year.
* Subjects with a history of true allergic response (ie, not intolerance) to more than one class of medications.
* Inability to tolerate oral medication or swallow tablets.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Reported Adverse Events (AEs) at 30 day Follow-Up | 30 day Follow-Up
Change from Baseline to Day 17 in Vital Signs | Baseline to Day 17
Change from Baseline to Day 17 ECGs | Baseline to Day 17
Change from Baseline to Day 17 Hematology | Baseline to Day 17
Change from Baseline to Day 14 Physical examination | Baseline to Day 14
Change from Baseline to Day 17 Body weight | Baseline to Day 17
Change from Baseline to Day 17 Serum chemistry | Baseline to Day 17
  Including Prolactin concentrations
Change from Baseline to Day 17 Urinalysis | Baseline to Day 17
Maximal peak steady-state plasma concentration | At Day 14
Minimum trough steady-state plasma concentration | At Day 14
Time to maximum peak steady-state plasma concentration | At Day 14
Area under the concentration-time curve during the dosing interval at steady-state | At Day 14
Terminal elimination half-life | At Day 14
For Brex only, apparent cleanse and apparent volume of distribution | At Day 14

SECONDARY OUTCOMES:
Mean change in CGI-S score | Day -1 of Dose Titration Phase to Day 7 and Day 14 of Fixed Dose Phase
Mean change in CGI-I score | Day 7 and Day 14
Glycosylated haemoglobin [HbA1c] | Baseline to Day 17
Change from Baseline to Day 17 Adrenocorticotropic hormone [ACTH] | Baseline to Day 17
Change from Baseline to Day 17 Cortisol | Baseline to Day 17
Change from Baseline to Day 17 Thyroid stimulating hormone [TSH] | Baseline to Day 17
Change from Baseline to Day 17 Prothrombin time [PT] | Baseline to Day 17
Change from Baseline to Day 17 Activated partial thromboplastin time [aPTT] | Baseline to Day 17
Change from Baseline to Day 17 International normalized ratio [INR] | Baseline to Day 17
For subjects with a current primary schizophrenia spectrum diagnosis, mean change in Positive and Negative Syndrom Scale (PANSS) | Day-1 to Day 15
For subjects with a current diagnosis of bipolar spectrum disorder, mean change in Young Mania Rating Scale (YMRS) | Day -1 to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization
Locations (10):
- United States (10):
  - Little Rock, Arkansas
  - Culver City, California
  - Orange, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Marlton, New Jersey
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - The Woodlands, Texas
  - Orem, Utah

IPD SHARING:
Plan to Share IPD: No